CLINICAL TRIAL: NCT01974505
Title: Learning Curve of Optiscope by Anesthesia Providers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jeju National University School of Medicine (Other)
Responsible Party: Principal Investigator, Hyun Jung Kim, Assistant professor, Jeju National University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: JejuNationalUniversityHospital
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Intubation, Intratracheal

ARMS (1):
- intubation using optiscope (Experimental): The investigators are novice on optiscope. They will perform intubation using optiscope to patients scheduled elective surgery.
  Interventions: Device: intubation using optiscope

INTERVENTIONS:
Device: intubation using optiscope — Optiscope (Clarus Medical, Minneapolis, MN, USA) is a semi-rigid fiberscope designed for endotracheal intubation. Anesthetic providers who are novice on optiscope will perform intubation using optiscope.

SUMMARY:
Optiscope (Clarus Medical, Minneapolis, MN, USA) is a semi-rigid fiberscope for endotracheal intubation. This study will investigate learning curve of Optiscope by anesthesia providers.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is scheduled general anesthesia for elective surgery

Exclusion Criteria:

* patient who is anticipated difficult airway
* patient who is needed rapid sequence induction
* Cervical injury

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
time to intubation | intubation period
  Time to intubation (from optiscope insertion to the detection of end tidal CO2) will be recorded. If time to inubation is longer than 180 s or pulse oxymetry is lower than 94%, mask ventilation will be performed. If intubation is not successful within 3 trials, it will be performed using direct laryngoscope.

CONTACTS AND LOCATIONS:
Locations (1):
- Jeju National University Hospital, Jeju City, Jeju Special Self-Governing Province, South Korea